CLINICAL TRIAL: NCT04428996
Title: Social Cognition and Interaction Training (SCIT) for Taiwanese People With Severe Mental Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-108-066
Record Dates: First submitted 2020-05-21; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Mental Health Disorder
Keywords: social cognition; Social cognition and interaction training; mental illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm AB (Experimental): "A" means SCIT program, and "B" means treatment as usual. Arm AB will receive a 60-minutes manual-guide SCIT session each week for 20 times first, then receive treatment as usual.
  Before the SCIT session, after the SCIT session and after 20 weeks treatment as usual, participants receive evaluations of clinical symptoms, emotional perception, theory of mind, and attributional bias.
  There are three main themes of the SCIT: 1) introduction and emotion, 2) figuring out situation and 3) integration: checking it out. After each theme of the intervention, participants will fill out a satisfaction survey.
  Interventions: Behavioral: Social Cognition and Interaction Training (SCIT)
- Arm BA (Experimental): "A" means SCIT program, and "B" means treatment as usual. Arm BA will first receive treatment as usual, then a 60-minutes manual-guide SCIT session each week for 20 times.
  At the first week, before and after the SCIT session, participants receive evaluations of clinical symptoms, emotional perception, theory of mind, and attributional bias.
  There are three main themes of the SCIT: 1) introduction and emotion, 2) figuring out situation and 3) integration: checking it out. After each theme of the intervention, participants will fill out a satisfaction survey.
  Interventions: Behavioral: Social Cognition and Interaction Training (SCIT)

INTERVENTIONS:
Behavioral: Social Cognition and Interaction Training (SCIT) — The social cognition and interaction training (SCIT) is a manual-guide group intervention that can apply to people with serious mental illness. There have been evidences showing that the SCIT could improve emotional perception, theory of mind, attribution bias, and social relationship.

SUMMARY:
Social cognition dysfunction (including emotional perception, theory of mind, and attribution bias) is a common dysfunction in serious mental illness, which may influence their life roles and daily functions. The social cognition and interaction training (SCIT) is a manual-guide group intervention that can apply to people with serious mental illness.Thus this study aims to conduct SCIT groups in Taiwan to investigate its feasibility and effectiveness.

This study will include 30 clients. Investigators will randomly allot participants into two group, and conduct a crossover design. The experimental group will receive a 60-minutes manual-guide SCIT session each week for 20 times, which will be leaded by 2 licensed occupational therapists. After the intervention, investigators will analyze demographic data and compare the difference between experimental group and control group on the social cognition performance.

DETAILED DESCRIPTION:
Social cognition dysfunction (including emotional perception, theory of mind, and attribution bias) is a common dysfunction in serious mental illness, which may influence their life roles and daily functions. The social cognition and interaction training (SCIT) is a manual-guide group intervention that can apply to people with serious mental illness. There have been evidences showing that the SCIT could improve emotional perception, theory of mind, attribution bias, and social relationship. However, there are no SCIT studies in Taiwan yet. Thus this study aims to conduct SCIT groups in Taiwan to investigate its feasibility and effectiveness.

This study will include 30 clients from a day care ward and community rehabilitation center, excluding clients with acute onset, brain injury, intellectual disability and substance abuse. The investigators will randomly allot participants into two group, and conduct a crossover design. Before and after the intervention protocol, both group receive evaluations of clinical symptoms, emotional perception, theory of mind, and attributional bias. The experimental group will receive a 60-minutes manual-guide SCIT session each week for 20 times, which will be leaded by 2 licensed occupational therapists. There are three main themes of the SCIT: 1) introduction and emotion, 2) figuring out situation and 3) integration: checking it out. After each theme of the intervention, participants will fill out a satisfaction survey. And a senior occupational therapist will observe the group and rate the fidelity of the group. The control group will receive treatment as usual.

After the intervention, the investigators will analyze demographic data and compare the difference between experimental group and control group on the social cognition performance.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mental illness

Exclusion Criteria:

* acute hospitalization within the past two months
* other diseases that may affect cognitive function, such as intellectual disability, substance abuse

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Test of Theory of mind #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  Includes language theory of mind and non-verbal theory of mind. Language theory of mind mainly measures the ability of cognitive components and emotional components. There are ten major questions, each of which contains four sub-questions. The first sub-question is a memory question, which must be answered correctly. The scores of the other three sub-questions are calculated. The full score of the language assignment is 30 points. There are ten questions in total, and the full score for non-verbal theory of mind is 20 points. About the internal consistency reliability, the language part is .91 and the non-verbal part is .93. About the test-retest reliability, the language part is .89 and the non-verbal part is .88.
Ambiguous Intentions Hostility Questionnaire #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  This is a measure of the attribution of the subject to the event, including 5 negative situations. Ask the subject to imagine that they are the protagonist in the situation. The first question responds to others' reasons for themselves. The second question is 6 The Likert scale (1 is absolutely not, 6 is absolutely yes) whether responding to others is intentional, the third question is to respond to your own with a 5 point Likert scale (1 is completely not, 5 is very angry) The degree of anger, the fourth question is also the degree of blaming others with a 5-point Likert scale (1 is not at all, 5 is absolutely), and finally asked the subjects to respond to the actions they will take; first Questions and the fifth question are evaluated by the evaluator based on his response. This is a tool with good reliability and validity, including internal consistency (alpha = .84 ~ .86) and inter-tester reliability (ICCs = .91 ~ .99).
Attributional Style Questionnaire #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  This is a questionnaire to assess the social cognition of the subjects, including the theory of mind, cognitive schema and verbal memory. There are 10 scenarios, each of which contains 3 yes-or-no questions, and one question is about degree of judgment. The scoring method is scoring according to three sub-items. The content of the response of the subjects is compared with the norm. If it is lower than two standard deviations, the degree is disabled.
Diagnostic Analysis of Nonverbal Accuracy, Taiwanese version #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  The DANVA-2-TW, a parallel version of the Diagnostic Analysis of Non-verbal Accuracy 2 (Nowicki and Duke, 1994), is a validated (Pan et al., 2009; Tseng et al., 2013), culturally suitable (Tseng et al., 2012) nonverbal measure for Han Chinese, considering that race and culture may considerably affect the accuracy of judging nonverbal emotions (Jack et al., 2012; Wickline et al., 2009). The DANVA-2-TW comprises 60 facial photographs and 60 voice clips representing specific emotions and intensities, including happy, sad, angry, fearful, and neutral stimuli.

SECONDARY OUTCOMES:
Self-Reported Graphic version of Personal and Social Performance rating scale #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  The PSP scale was developed for assessing patients' function by mental health professions . The rater can assess one global score as well as sub-scores of the four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviors. The PSP showed good interrater (ICC = 0.87) and test-retest (ICCs > 0.90) reliability (Patrick et al., 2009) and adequate validity (Cronbach aloha = 0.76) (Kawata & Revicki, 2008). As many studies showed that people with schizophrenia have greater impairment in processing speed and verbal memory than visual spatial-perception memory, a graphic version of PSP (SRG-PSP) was developed. The results of this SRG-PSP were significantly correlated to those of their corresponding criteria on the PSP. The SRG-PSP total score ranges from 12 to 51, and the higher the score, the better social performance.
Trail Making Test #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  This is a test to assess visual attention, task conversion, processing speed and cognitive flexibility. Contains two parts. Part A is a number from 1-25, and the subjects must connect the numbers in order. Part B contains 12 numbers and 12 letters. The subjects must connect the numbers and the zodiac in sequence (1-Mouse-2-Bull-3 ...). The scoring method is the individual seconds to complete these two tasks. According to the research by Wang et al. In 2018, this tool has good reliability (ICC> .75).

OTHER OUTCOMES:
Brief Psychiatric Rating Scale | baseline
  The BPRS (Overall & Gorham, 1962) is one of the most frequently used instruments for evaluating psychopathology in people with schizophrenia. Its psychometric properties in terms of reliability, validity and sensitivity have been extensively examined (Leucht et al., 2005). It measures psychiatric symptoms such as depression, anxiety, hallucinations and unusual behavior. Each symptom is rated 1 (not present) to 7 (extremely severe).
Brief Symptom Rating Scale-50 #Change from baseline at 20 weeks and 40 weeks | baseline, 20th week, 40th week
  Lee, Lee, Yen, Lin, and Lue (1990) revised the Symptom Checklist-90-R scale (Derogatis, Rickels, & Rock, 1976) to develop BSRS-50. The scale contains 50 symptom descriptions and can be summarized into 10 concepts, including physicalization, compulsiveness, interpersonal sensitivity, depression, anxiety, hostility, fear, suspiciousness, psychosis and additional symptoms. Subjects report the degree of distress they feel based on each symptom. Each item is rated 0-4 points, 0 points: no, 4 points: very powerful. Research supports BRSR-50 with good psychometric characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Yi chia Liu, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No